CLINICAL TRIAL: NCT03221855
Title: Randomized Clinical Trial: Use of Domperidone to Increase Milk Production in Mothers With Newborns Hospitalized in Neonatology
Brief Title: Use of Domperidone to Increase Milk Production in Mothers With Newborns in Neonatology
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-0197
Record Dates: First submitted 2016-09-16; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Domperidone; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Domperidone (Active Comparator): Domperidone 10mg every 8 hours for 7 days.
  Interventions: Drug: Domperidone
- Placebo (Placebo Comparator): Placebo 10mg every 8 hours for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Domperidone — Capsules 10mg orally each 8 hours for 7 days.
  Other Names: Motilium
  Arms: Domperidone
Drug: Placebo — Capsules 10mg orally each 8 hours for 7 days.
  Other Names: Lactose capsules
  Arms: Placebo

SUMMARY:
It is a double-blind randomized clinical trial placebo-controlled, which aims to assess whether Domperidone medication helps to increase milk production. The sample of 30 mothers of newborns in the Neonatal Intensive Care Unit of the Hospital de Clínicas de Porto Alegre for at least 15 days, receiving power enteral tube (without clinical condition for oral). Nursing mothers will be evaluated by the researcher (breastfeeding committee member) or consultants in breastfeeding that will advise these women about the practice of runs out of the breasts each mother. You receive containers for collection, at least one for each time you run out. These containers will measure the volume of milk. For each mother that refer insufficient milk production or is not maintaining adequate production for their newborn within 24 hours, one will be generated data form and after 15 days postpartum will be randomized and receive domperidone orally at a dose of 10mg 8/8 hours, or placebo in same volume. The milk volume will be measured daily. Three blood samples will be collected for each lactating each with 5 ml tube without anticoagulant for analysis of serum prolactin and domperidone. The sample 01 will be collected immediately after randomization, before receiving any medication (placebo x domperidone). The sample 02 on 5 of the study. And the sample 03, day 10 of the study, three days after the termination of the use of medication or placebo. A milk sample (5 ml) of each mother will be collected on day 5 to analysis of domperidone levels in milk. Once collected, the samples will be processed and frozen at -80o C for later analysis. All mothers will be followed until hospital discharge of their newborns, to monitor outcome breastfeeding exclusive breast.

DETAILED DESCRIPTION:
It is a clinical double-blind randomized placebo-controlled trial. The sample consists of 30 mothers of newborns stable hemodynamically and are admitted to the Neonatal Intensive Care Unit of the Hospital de Clínicas de Porto Alegre for at least 15 days, receiving power via enteral tube (without clinical condition to oral). The mothers will be assessed by the researcher (committee member of breastfeeding) or a lactation consultants who will advise women about these practice runs out of the breasts. Breast milk is collected using a breast pump electric Lactinadouble, which enables the extraction of milk in both breasts simultaneously. Every mother receive collection containers, at least one for every time you run out. These containers will measure accurately the volume of milk. Women will be instructed to use a new packaging for each pumping and not add the milk from two different milkings. For every mother noted that insufficient milk supply or production is not suitable for keeping your newborn within 24 hours, it will generate an data form and after 15 days postpartum will be randomized and receive domperidone orally at a dose of 10mg of 8/8 hours or placebo in same volume. The mothers included in the survey will receive record sheets and adhesive labels to record the amount of milk collected, the date and time. The milk volume will be measured daily. Three blood samples will be collected for each nurse, each with 5 ml tube analysis without anticoagulant for serum levels of prolactin and domperidone. The sample 01 will be collected immediately after randomization, before receiving any medication (placebo x domperidone). The sample 02 at day 5 of the study. And the sample 03, the 10th day of the study, 3 days after the end of the medication or placebo.A milk sample (5 ml) of each mother will be collected on day 5 to analyzing levels of domperidone in the milk. Once collected, the samples will be processed and frozen at-80o C for later analysis. All mothers will be followed until discharge of their newborns, to monitor outcome breastfeeding exclusive breast.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who report a decrease in the production of depleted milk.
* Mothers who do not have sufficient milk production to supply the baby's demand, according to the amount prescribed in the medical prescription.
* Mothers who are able to swallow tablets.

Exclusion Criteria:

-Mothers with the virus HIV.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Increase the production of breast milk of nursing mothers who are with their newborns admitted to the neonatal. Milk production measured by volume (ml) for 10 days. | 10 days
  Increase the production of breast milk of nursing mothers who are with their newborns admitted to the neonatal, failing to provide this Baby breastfed during their hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Rita de Cassia C. Silveira, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Giugliani ER. [Breast-feeding in clinical practice]. J Pediatr (Rio J). 2000 Nov;76 Suppl 3:S238-52. doi: 10.2223/jped.161. Portuguese. PMID 14676902
- [Background] Charpak N, Ruiz-Pelaez JG, Figueroa de C Z, Charpak Y. A randomized, controlled trial of kangaroo mother care: results of follow-up at 1 year of corrected age. Pediatrics. 2001 Nov;108(5):1072-9. doi: 10.1542/peds.108.5.1072. PMID 11694683
- [Background] Zuppa AA, Sindico P, Orchi C, Carducci C, Cardiello V, Romagnoli C. Safety and efficacy of galactogogues: substances that induce, maintain and increase breast milk production. J Pharm Pharm Sci. 2010;13(2):162-74. doi: 10.18433/j3ds3r. PMID 20816003
- [Background] Gabay MP. Galactogogues: medications that induce lactation. J Hum Lact. 2002 Aug;18(3):274-9. doi: 10.1177/089033440201800311. PMID 12192964
- [Background] Anderson PO, Valdes V. A critical review of pharmaceutical galactagogues. Breastfeed Med. 2007 Dec;2(4):229-42. doi: 10.1089/bfm.2007.0013. PMID 18081460
- [Background] da Silva OP, Knoppert DC, Angelini MM, Forret PA. Effect of domperidone on milk production in mothers of premature newborns: a randomized, double-blind, placebo-controlled trial. CMAJ. 2001 Jan 9;164(1):17-21. PMID 11202662
- [Background] Wan EW, Davey K, Page-Sharp M, Hartmann PE, Simmer K, Ilett KF. Dose-effect study of domperidone as a galactagogue in preterm mothers with insufficient milk supply, and its transfer into milk. Br J Clin Pharmacol. 2008 Aug;66(2):283-9. doi: 10.1111/j.1365-2125.2008.03207.x. Epub 2008 Apr 21. PMID 18507654
- [Background] Djeddi D, Kongolo G, Lefaix C, Mounard J, Leke A. Effect of domperidone on QT interval in neonates. J Pediatr. 2008 Nov;153(5):663-6. doi: 10.1016/j.jpeds.2008.05.013. Epub 2008 Jun 27. PMID 18589449
- [Background] Campbell-Yeo ML, Allen AC, Joseph KS, Ledwidge JM, Caddell K, Allen VM, Dooley KC. Effect of domperidone on the composition of preterm human breast milk. Pediatrics. 2010 Jan;125(1):e107-14. doi: 10.1542/peds.2008-3441. Epub 2009 Dec 14. PMID 20008425
- [Background] Zavitsanos AP, MacDonald C, Bassoo E, Gopaul D. Determination of domperidone in human serum and human breast milk by high-performance liquid chromatography-electrospray mass spectrometry. J Chromatogr B Biomed Sci Appl. 1999 Jun 25;730(1):9-24. doi: 10.1016/s0378-4347(99)00163-2. PMID 10437667